CLINICAL TRIAL: NCT06952231
Title: Comparison of Effect of Sitagliptin and Empagliflozin in Combination With Metformin on High-Sensitivity C-Reactive Protein Levels in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Sitagliptin and Empagliflozin in Combination With Metformin on Hs-CRP Levels in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Lahore (Other)
Collaborators: University of Lahore Hospital (ULH) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ERC1212311
Record Dates: First submitted 2025-03-27; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate; Metformin; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Sitagliptin (as phosphate monohydrate) 50 mg twice daily plus metformin HCl 1000 mg twice daily
  Interventions: Drug: Sitagliptin + Metformin
- Group B (Active Comparator): Empagliflozin 12.5 mg twice daily plus metformin HCl 1000 mg twice daily
  Interventions: Drug: Empagliflozin + Metformin

INTERVENTIONS:
Drug: Sitagliptin + Metformin — Self administration of Sitagliptin (as phosphate monohydrate) 50 mg twice daily plus metformin HCl 1000 mg twice daily
  Arms: Group A
Drug: Empagliflozin + Metformin — Self administration of Empagliflozin 12.5 mg twice daily plus metformin HCl 1000 mg twice daily.
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to compare the effects of Sitagliptin and Empagliflozin in combination with metformin on High sensitivity C reactive proteins (hs-CRP) levels and efficacy in T2DM patients.

The main question aims to answer are the difference in effect of Sitagliptin with metformin and Empagliflozin with metformin on the levels of hs-CRP, HbA1C, Fasting blood glucose and BMI in patients with type 2 diabetes millitis.

The sample size for the trial is 25 participants in each group based on 95% level of confidence and 80% power of the study.

Fifty participants fulfilling the eligibility criteria will be randomly divided into two groups

* Group A will be taking sitagliptin 50 mg along with metformin 1000mg BD for 12 weeks and group B will be taking Empagliflozin 12.5mg along with metformin 50mg for 12 weeks.
* They will visit the hospital fortnightly for check up for 1st month and then monthly for tests
* Participants will keep the record of their fasting blood glucose levels and any adverse effects during course of study.

Primary outcomes measures: hs-CRP Secondary outcome measures: HbA1c, fasting blood glucose (FBG), body mass index (BMI).

DETAILED DESCRIPTION:
INTRODUCTION The worldwide prevalence of diabetes is high and continues to rise, with a projected increase of 84% across South East Asia by 2045. Pakistan ranks third in the world with 30.8% of adults having diabetes and is expected to have the highest prevalence if current trends continue. According to American Diabetic Association (ADA), Metformin is the 1st line pharmacological treatment for type 2 diabetes mellitus (T2DM). Unfortunately, the majority of patients who initially attain glycemic control with metformin do not sustain adequate glycemic control over the long term and require an additional antidiabetic agent. Sitagliptin (a dipeptidyl peptidase-4 inhibitor) and Empagliflozin (Sodium glucose-cotransporter 2 inhibitor) are considered as effective and safe metformin adjuncts.

Cardiovascular diseases are known complications in individuals with T2DM. The newer antiglycemic agents are acknowledged for their ability to offer cardiovascular advantages in addition to facilitating improved glycemic control. The underlying mechanism most likely associated with these cardiovascular benefits is closely linked to their anti-inflammatory properties. It is well-established that inflammatory markers tend to escalate in the presence of diabetes. Among other inflammatory markers, the high-sensitivity C-reactive protein (hs-CRP) serves as a reliable indicator for the development of cardiovascular disease among individuals diagnosed with diabetes.8 It is synthesized by the liver and increases during acute responses to infection or tissue damage. Drugs that effectively reduce hs-CRP inhibit atherosclerosis progress, especially in patients with diabetes.

Previous researches showed that sitagliptin and empagliflozin reduce inflammation in diabetic patients with known cardiovascular risk factors. According to a previous study, the mean reduction in hs-CRP from base line in sitagliptin plus metformin and sulfonylurea group was 0.53±0.26 and in pioglitazone plus metformin and sulfonylurea group, was 2.44±0.20. Both groups had statistically significant difference in these values (p-value = 0.04). Another study showed the significant decrease that is 0.59±0.42 in hs-CRP levels by empagliflozin alone as compared to placebo.

Despite the availability of studies on effect of some antiglycemic agents on hs-CRP levels, there is a lack of scientific data comparing the effects of sitagliptin and empagliflozin as add-ons to metformin in reducing C-reactive protein levels in diabetic patients without cardiovascular diseases. Additionally, no studies have been found in our country comparing the effects of these combinations on C-reactive protein levels in diabetic patients. This study aims to compare the effect of sitagliptin and empagliflozin in combination with metformin on hs-C reactive protein levels in patients with T2DM.

This study will help in providing better management guideline for prevention of cardiovascular complications among patients having Type 2 diabetes mellitus.

OBJECTIVES:

To compare the effect of sitagliptin and empagliflozin in combination with metformin on hs-C reactive protein levels in patients with T2DM.

OPERATIONAL DEFINITIONS:

1. Type-2 Diabetes:

   Patient having type 2 diabetes mellitus (T2DM) when he/she has i. Fasting blood glucose (FBG) level ≥ 7.0 mmols/L ii. HbA1 c ≥ 6.5%
2. Hs-CRP: Hs-CRP levels are the amount of C-reactive protein, a marker of inflammation, in the blood as measured by Enzyme-linked Immunosorbent Assay (ELISA) method. Normal levels are <1.0 mg/L.

ALTERNATE HYPOTHESIS:

There is a difference in pre and post hs-CRP level among three interventional groups

MAIN OUTCOMEE MEASURES:

Primary outcomes measures: hs-CRP Secondary outcome measures: HbA1c, fasting blood glucose (FBG), body mass index (BMI)

MATERIAL AND METHODS:

Study design: Prospective Cohort study Setting: University of Lahore Teaching Hospital (ULTH), The University of Lahore (UOL), Lahore Duration of study: 12 months Sampling size: Calculated through WHO software for comparison of means Margin of error =5% Confidence level=95% Power of test= 80%. Population SD: 1.2 Population variance: 1.44 The anticipated means ± SD of hs-CRP is 0.53±0.2611 in sitagliptin plus metformin group vs 0.59±0.4212 empagliflozin plus metformin group.

Sample size in each group = 25 patients Total sample size= 50 Sampling technique: It will be non probability, consecutive sampling

Sample Selection:

Inclusion criteria:

Type 2 diabetes patients aged ≥18, both genders, who were taking Metformin ≥ 1000 mg daily since 1 year.

Exclusion criteria:

The following patients will be excluded from the study i. Patients with type 1 diabetes mellitus ii. Patients with acute systemic infections (tonsillitis, chest infections, UTI, Gynecological infections) on the basis of history, examination and ancillary investigations when necessary.

iii. Patients with history of malignancy, angina and myocardial infarction, thyroid problems.

iv. Patients with liver disease/renal disease/ deranged liver function tests and renal function tests will be excluded from the study v. Pregnancy, lactation.

Patients and Methods:

A total of 50 patients will be enrolled in the study after obtaining informed and written consent. The patients will be randomly assigned into three groups namely A and B each comprising of 25 patients. The objectives, procedure and possible complications will be explained to each study participant. Each group will be given the study drug in consultation with senior faculty member (diabetologist) of medicine department of ULTH as follows.

Group A (n=25): Sitagliptin (as phosphate monohydrate) 50 mg twice daily plus metformin HCl 1000 mg twice daily Group B(n=25): Empagliflozin 12.5 mg twice daily plus metformin HCl 1000 mg twice daily.

The patients will be called for follow up at fortnightly interval. Each patient will be assigned a code and visit date will be recorded accordingly. The patient will be advised to report principal investigator immediately in case of any adverse event including hypoglycemia. The treatment protocol will be discontinued in the following cases:

i. Acute allergic reactions to any of the drug. ii. Specific toxic effects suspected on the basis of history and examination and confirmed by investigations where necessary.

iii. Patient not willing to follow or participate the study protocol. The renal and hepatic profile will be checked at the time of screening and in case patient was found to have deranged hepatic or renal profile, he/she will be excluded from the study.

This study will be conducted in conformity with the approval of the ethical committee of the institution. The study will also adhere to Good Clinical Practice guidelines13 and follow principles outlined by the World Medical Association's Helsinki Declaration.14

DATA COLLECTION PROCEDURE:

A predesigned proforma will be used to collect the information regarding the date of screening, patient bio-data profile, record of study parameters, discontinuation of treatment protocol and any adverse event related to study procedures.

The baseline hs-CRP and FBS, HbA1c will be determined by taking a blood sample of 5 ml taken using aseptic measures on day zero. Hs-CRP and FBS will be measured at 4, 8 and 12 weeks while the HbA1c will be measured after 12 weeks. Confidentiality of the data will be ensured.

DATA ANALYSIS PROCEDURE:

Data will be entered on SPSS- software version 23 with age, hs-CRP, FBG, BMI as numeric variables and gender as categorical variables. Comparison between CRP levels will be made using one-way ANOVA and significance will be tested at p-value of 0.05. Qualitative data will be presented in the form of frequencies and percentages. The quantitative variables will be described by mean and standard deviation. Graphs will be used for data visualization. Post hoc Tukey's test will be used for intergroup comparisons at different times. Paired t-test will be used for intragroup comparisons at different times.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients aged ≥18, both genders, who were taking Metformin ≥ 1000 mg daily since 1 year.

Exclusion Criteria:

* Patients with acute systemic infections (tonsillitis, chest infections, UTI, Gynecological infections) on the basis of history, examination and ancillary investigations when necessary. Patients with history of malignancy, angina and myocardial infarction, thyroid problems, Patients with liver disease/renal disease/ deranged liver function tests and renal function tests will be excluded from the study, Pregnancy, lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
hs-CRP | 12 weeks
  Difference in levels of hs-CRP before intervention and 4, 8 and 12 weeks of intervention

SECONDARY OUTCOMES:
HbA1C | 12 weeks
  The quantitative levels of HbA1c
Fasting Blood Glucose | 12 weeks
  Self detection of fasting blood glucose levels
Body mass index (BMI) | 12 weeks
  Calculation of BMI on a numerical scale

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No